CLINICAL TRIAL: NCT02143219
Title: Phase-2 Study Evaluating Overall Response Rate (Efficacy) and Autonomy Daily Living Preservation (Tolerance) of "FOLFIRINOX " Pharmacogenetic Dose Adjusted, in Elderly Patients (70 yo. or Older) With a Metastatic Pancreatic Adenocarcinoma.
Brief Title: Efficacy and Tolerance Evaluation in FOLFIRINOX Dose Adjusted in Elderly Patients With a Metastatic Pancreatic Cancer
Acronym: PAMELA70
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICO-N-2014-01; 2014-000539-17 (EudraCT Number)
Record Dates: First submitted 2014-05-14; First posted 2014-05-21 (Estimated); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Pancreatic Metastatic Cancer; Toxicity
Keywords: Pancreatic metastatic cancer; FOLFIRINOX; toxicity; efficacy
MeSH Terms: interventions — Oxaliplatin; Leucovorin; Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FOLFIRINOX (Other): FOLFIRINOX (D1-D15, for maximum 12 cycles) = Oxaliplatine + Folinic acid + Irinotecan + 5-FU
  Interventions: Drug: Oxaliplatine; Drug: Folinic acid; Drug: Irinotecan; Drug: 5-FU

INTERVENTIONS:
Drug: Oxaliplatine — Oxaliplatine : 85mg/m², 2-hours IV infusion (D1),
  Other Names: Eloxatine®
Drug: Folinic acid — Folinic acid (FA): 400 mg/m² , 2-hour IV infusion (D1),
Drug: Irinotecan — Irinotecan (at the dosage determined by the UGT1A1 status), 90 min IV infusion starting 30 min after the FA starts
  * Homozygous 6/6 or 6/7: irinotecan will start at 150 mg/m², then will be increased according to clinical/biological tolerance by 10% steps, at each cycle, up to 180 mg/m² at max.
  * Homozygous 7/7: irinotecan will start at 130 mg/m² in the first cycle then be increased up to a max of 150 mg/m², by 10% steps, according to tolerance.
  Other Names: Campto®
Drug: 5-FU — 5-FU (according to the DPD pharmacogenetic status), continuous IV infusion of 46 hours, starting at the end of FA infusion:
  * If no DPD deficiency, 5-FU start at 1600 mg/m² and can be modulated according to clinical/biological tolerance after each course, i.e., 1800 mg/m² the 2nd course and 2000 mg/m² the 3rd one
  * If partial DPD deficiency: 5-FU start at 1200 mg/m² and can be increased up to 1800, then 2000 if the clinical/biological tolerance are good at the 2nd and 3rd course.
  Other Names: 5-fluorouracile

SUMMARY:
Metastatic pancreatic carcinomas represent the 5th cause of cancer death in France (#8000 per year). The median age at diagnosis is 69 and 74 in male and female respectively. When the 5-Fluorouracile has been used as a single agent with a limited efficacy during more than 20 years, the onset of gemcitabine in 1995 has led to a moderate increase of median survival (from 4.41 to 5.65 months) and overall survival at 1 year (2 versus 18%). Recently, in a phase II followed by a phase-III study, a French collaborative group has demonstrated the benefit of "FOLFIRINOX " regimen versus gemcitabine alone, in terms of median survival (11.1 versus 6.8 months), progression-free survival (6.4 versus 3.3 months) and response rate (31.6 versus 9.4%).

Although more hematologic (neutropenia) and GI toxicities were observed, FOLFIRINOX was acceptable as a new standard regimen for the majority of patients under the age of 70 with a good Performans Status. To reduce the toxicity of FOLFIRINOX in elderly patients (> 70 yo), pharmacogenetic monitoring of 5-FU and Irinotecan key metabolism enzymes (DPD and UGTA1) may be easily performed. The methodology of the study is to use the Bryant & Day statistical method, allowing to consider simultaneously as principal objective, the response rate (efficacy) and the tolerance (preservation of autonomy daily living, Katz index): this design is particularly fitting in a study for elderly patients who represent half of the pancreatic carcinoma population.

DETAILED DESCRIPTION:
METHODOLOGY :

Phase II study, opened, multicentric

MAIN OBJECTIVE :

The main objective is the simultaneous evaluation of the objective rate of answer and toxicity of her(it) of the protocol FOLFIRINOX administered to doses adapted at patients of 70 and more years old.

SECONDARY OBJECTIVE :

* Efficiency evaluation;
* Tolerance evaluation;
* Quality of Life (QoL) and clinical profit.

STATISTICAL ANALYSIS:

An analysis in two stages is planned, according to the method of Bryant and Day with a risk ß 5 % to reject wrongly an effective treatment and of acceptable toxicity and a risk a=10 % to accept wrongly a not rather effective or too toxic treatment.

The study will be considered as successful if:

* we obtain at least 11 tumoral answers and
* maxi 30 patients on 72 are in loss of autonomy (decrease of their ADL).

  * All the patients who will have received at least an injection will be eligible for the evaluation of the toxicity
  * The evaluation of the efficiency will be made after 3 cures at least unless early termination where the scanner will be anticipated.
  * All the toxicity will be increased according to criteria of toxicity NCI-CTC v4.0.
  * The evaluation of the tumoral answer (CR, PR and SD) will be made according to the criteria RECIST-v1.1.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven ductal pancreatic carcinoma
* Metastatic disease
* First-line treatment : No previous chemotherapy in metastatic stage but adjuvant treatment before relapse (secondary metastatic) is permitted, provide it has been administered more than 6 months before)
* Age of 70 yo or above
* Normal DPD enzyme level or partial defect (excluding total defect)
* Adequate bone marrow reserve: as indicated by : neutrophils >1500/mm3, platelets >100,000/ mm3, Hb >10.0g/dL.
* Adequate Renal function as indicated by: MDRD creatinine clearance > 50ml/min.
* Adequate hepatic function as indicated by: serum bilirubin < 1.5 times the upper limit of normal, AST and ALT < 2.5 times the upper limit of normal, or < 5 times the upper limit of normal if liver metastases are present.
* Written informed consent must be obtained prior to protocol-specific procedures are being performed
* Patient is affiliated to a social security category

Exclusion Criteria:

* Other than ductal pancreatic carcinoma: namely endocrin tumors, acinar cells carcinoma, cystadenocarcinoma or adenocarcinoma of the ampulla of vater
* Non-metastatic but locally advanced pancreatic adenocarcinoma
* Complete DPD deficiency
* History of Cardiac failure or symptomatic coronary artery disease
* Autonomy Daily Living score by Katz <4
* Prior treatment with FOLFIRINOX (adjuvant)
* Major comorbidity likely to be an obstacle to treatment
* Active or uncontrolled infection such as HIV or chronic B or C hepatitis
* Uncontrolled diabetes mellitus
* Prior peripheral neuropathy, grade > 2
* Inflammatory bowel disease localized on the colon or rectum; bowel obstruction or severe uncontrolled diarrhea
* Previous or concomitant malignancies other than effectively treated carcinoma in situ of the cervix or non-melanoma skin cancer
* Hereditary fructose intolerance
* Persons deprived of liberty or under guardianship
* Any social, geographical or psychological condition which would compromise the ability to fully comply with the trial procedures and treatments

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-07-31 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
1st step analysis : Safety and efficacy after 34 patients included | 12 weeks after the 34th patient included
  Evaluation of Efficacy: Progression-free-Survival (PFS) and Overall Survival (OS) will be evaluated.
  Evaluation of Toxicity: Will be analyzed, according to the NCI-CTCAE version 4.0:
  * The incidence of hematological toxicities (grade 3-4, in particular neutropenia and febrile neutropenia)
  * The incidence of GI toxicities, in particular diarrhea and oral mucositis
  * The incidence of peripheral neuropathies
  For statistical analysis :
  either >= 17 patients show a decrease of their ADL (of 1.5 ADL or more) : the treatment is considered as being too toxic, either <= 3 patients presented a tumoral response: the treatment is considered as not being effective enough,
  => The study will then be arrested in this 1st stage.

SECONDARY OUTCOMES:
2nd step analysis : Safety and efficacy after 72patients included | 12 weeks after the 72th patient included
  Only if 1st step is successful we can do the second step :
  * For toxicity : if >= 31patients show a decrease of their ADL (of 1.5 ADL or more) and/or
  * For efficacy : if <= 10 patients presented a tumoral response
    => Study is successful if :
  * we obtain at least 11 tumoral response and
  * maximum 30 patients on 72 evaluable are in loss of autonomy (ADL)

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine HIRET, MD, Principal Investigator — Institut de Cancérologie de l'Ouest (ICO) - Nantes, France
Locations (6):
- France (6):
  - ICO Paul Papin, Angers
  - CH Vendée, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille
  - ICM (Val d'Aurelle), Montpellier
  - Centre Eugène marquis, Rennes
  - ICO René Gauducheau, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No